CLINICAL TRIAL: NCT06037902
Title: Use of CPAP (Continuous Positive Airway Pressure) for Simulating Esophageal Cancer Patients Prior to Radiotherapy
Brief Title: CPAP for Esophageal Cancer With Radiotherapy
Acronym: TROS-7
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Yaacov Lawrence, Chair of Department of Radiation Oncology, principal investigator, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-22-0032-YL-CTIL
Record Dates: First submitted 2023-08-28; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Esophageal Cancer
Keywords: radiation
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: all patients undergo two simulations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CPAP (Experimental): patients will undergo simulation twice, with and without CPAP
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — patients undergo simulation twice, with and without CPAP

SUMMARY:
The goal of this clinical trial is to test the use of CPAP in patients with esophgaeal cancer undergoing radiotherapy.

The main questions it aims to answer are:

* does use of CPAP decrease exposure of normal lung to radiation?
* does use of CPAP decrease exposure of normal heart to radiation?

Participants will undergo simulation twice:

* with CPAP
* without CPAP

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cancer, with a tumor (primary or secondary) in the esophagus including tumors in the esophagus-stomach junction.
2. Age ≥ 18
3. Planned RT treatment
4. The level of functioning ≥ 60 on the Karnofsky scale
5. Life expectancy ≥ two months
6. All patients must understand the informed consent form document and sign it of their own free will before any test/procedure related to the study is performed.
7. Able to undergo simulation and radiation with CPAP
8. Candidate patients can be recruited to receive definitive, palliative or pre-operative radiation, with or without chemotherapy.

Exclusion Criteria:

A person who meets any of the following exclusion criteria will not be able to participate in the study:

1. Pregnancy or breastfeeding
2. Significant comorbidity at the starting point that would prevent the use of CPAP
3. Hospitalized in an institution by virtue of an administrative order or a court order.
4. Special population
5. A history of a psychiatric problem that may impair the patient's ability to understand the research requirements or respond to them, or to give his consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
absolute mean heart radiation dose | on day of simulation (day 1)
  measured in Gy

SECONDARY OUTCOMES:
lung dose in Gy | on day of simulation (day 1)
  mean lung dose, V5 and V20
heart dose in Gy | on day of simulation (day 1)
  mean heart dose, V30
movement of tumor in cm | on day of simulation (day 1)
  how much tumor moves with breathing

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No